CLINICAL TRIAL: NCT04257695
Title: Developing and Pilot Testing an Intervention to Increase Opioid Tapering in Primary Care
Brief Title: Developing and Pilot Testing an Opioid Tapering Protocol
Acronym: TapPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Hector Perez, Principal Investigator, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-10910; K23DA044327 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Chronic Pain; Opioid Use; Analgesia
Keywords: opioid; tapering; chronic pain
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TapPro (Experimental): Biweekly telephone and in-person visits with a clinician over three months. At each visit, a protocol adapted from the Prescription Opioid Taper Study will be provided to participants, who will learn about pain coping, distraction techniques, diaphragmatic breathing, sleep techniques, and progressive muscle relaxation techniques. All are specifically designed for patients with chronic pain on chronic opioid therapy. During visits, taper parameters will be discussed and the provider will work through a dose reduction schedule, if participants are in agreement. Additionally, urine drug screens will be obtained.
  Interventions: Behavioral: TapPro
- Usual Care (No Intervention): Participants randomized to the usual care arm will continue seeing their primary care providers as indicated.

INTERVENTIONS:
Behavioral: TapPro — Manualized intervention administered by a clinician to facilitate opioid tapering during clinical visits.
  Arms: TapPro

SUMMARY:
This study proposes to pilot test an intervention to facilitate opioid pain reliever (OPR) tapering in primary care. The intervention will incorporate a clinician embedded within primary care to follow tapering dose schedules to support providers as well to deliver a psychosocial curriculum to support and engage patients. In a pilot randomized controlled trial (RCT), the study will examine the preliminary efficacy and feasibility of the manualized, protocol-based tapering intervention ("TapPro") compared to usual care. As there is no standard definition or outcome for tapering, the primary efficacy outcome is a decrease in OPR dose over six months. Separately, the study proposes a clinically meaningful dose reduction (greater than or equal to 30 percent) as a secondary outcome. The central hypotheses' are that a tapering intervention with patient and provider support is feasible in a primary care setting and can result in greater dose reduction when compared to usual care.

DETAILED DESCRIPTION:
In a 12-week randomized controlled trial based in a primary care outpatient clinic, the study will recruit 60 patients on moderate to high dose chronic opioid therapy for whom providers recommend opioid tapering and randomize 1:1 to an opioid tapering protocolized intervention (TapPro) or to usual care. Over three months, participants in the TapPro arm will visit with a clinician on the telephone on a biweekly basis in order to facilitate opioid prescribing and tapering and a pain self-care and coping curriculum. In the control arm, participants will see their primary care providers as per usual and decisions on opioid prescribing and tapering will be made by the primary care providers. Participants will be assessed throughout the study with questionnaires, urine drug screens, prescription database review, and medical record review.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18
2. chronic prescription opioid use (>3 monthly prescriptions from the clinic within prior 6 months)
3. morphine milligram equivalents (MME) ≥50
4. poorly controlled pain (PEG pain score ≥ 5/10)
5. providers considering opioid taper but no reductions in opioid dose over the past 6 months.

Exclusion Criteria:

1. Active cancer or other serious progressive illness, by medical review and by self-report
2. Moderate or severe opioid use disorder, as per DSM-V
3. Inability to give informed consent
4. Active suicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in opioid dose over six months | Up to six months
  Repeated measure analysis of opioid dosage over six months

SECONDARY OUTCOMES:
Opioid dose reduction | Up to six months
  Dichotomous outcome assessing whether participant reached a thirty percent or greater opioid dose reduction
Patient reported pain score | Up to six months
  Repeated measure analysis of pain severity, as per the PEG pain screening tool. The PEG is a 3 item scale that assesses pain intensity and interference on a 0 to 10 scale where 0 equals "no pain" and 10 is "pain as bad as you can imagine"
Pain interference | Up to six months
  Repeated measures analysis of pain interference, as per the Brief Pain Inventory (BPI) pain interference subscale. The BPI pain interference subscale is scored as the mean of 7 interference items, scored from 0 (does not interfere) to 10 (completely interferes).
Pain related self-efficacy | Up to six months
  Repeated measures analysis of pain related self-efficacy, as per the Pain Self-Efficacy Scale. The Pain Self-Efficacy scale consists of 10 questions that assess a patient's confidence in performing tasks in spite of pain. It is scored from 0 (not at all confident) to 6 (completely confident). Higher scores are better.
Change in Quality of life score | Up to six months
  Repeated measures analysis of two different quality of life scores, as per the EQ-5D and the Assessment of Quality of Life 8-item scale (AQoL-8D). The EQ-5D measures quality of life in 5 different domains in 5 questions. The AQoL-8D measures quality of life in 8 different domains in 35 questions. Higher scores denote greater quality of life.
Depressive symptoms | Up to six months
  Repeated measures analysis of depression scores, as per the Center for Epidemiologic Studies Depression Scale (CES-D). This is a 20 item questionnaire that assesses the frequency of several depressive symptoms, rated from 0 (rarely or none of the time) to 3 (most or all of the time). Lower scores mean fewer depressive symptoms.
Anxiety symptoms | Up to six months
  Repeated measures analysis of anxiety scores, as per the Brief symptom anxiety subscale. This is a 40 item questionnaire that assesses the frequency of symptoms of anxiety. It is scored from 1 (almost never) to 4 (almost always). Lower scores mean less anxiety.
Pain catastrophizing | Up to six months
  Repeated measures analysis of the Pain Catastrophizing Scale. This is a 13 item scale scored from 0 (not at all) to 4 (all the time) about symptoms associated with pain catastrophizing. Lower scores denote less pain catastrophizing.
Sleep quality | Up to six months
  Repeated measures analysis of sleep quality, as per the Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-ME) Sleep Impact Short Form. This is a 5 item survey of sleep symptoms, scored from 1 (always) to 5 (never), with higher scores meaning more problems with sleep.
Opioid Misuse | Up to six months
  Repeated measures analysis of opioid misuse, as per the Current Opioid Misuse Measure (COMM) score. It is a 17 item survey, rated from 0 (never) to 4 (very often), assessing behaviors associated with opioid misuse. Higher scores are associated with greater opioid misuse.
Opioid Knowledge | Up to six months
  Change in Opioid Knowledge score, as per the Survey for Pain Attitudes, Knowledge, and Beliefs (SOPA+KB). This is an 18 question survey that assesses agreement with several pain statements, rated from 1 (do not agree) to 4 (completely agree). Higher scores denote better knowledge.

OTHER OUTCOMES:
Retention in care | 12 months
  Dichotomous outcome -more than or equal to 1 visit with primary care physician (PCP) during six month study period AND more than or equal to 1 visit with PCP during next six months
Percent of patients attending clinic visits | 6 months
  Percent of patients who attend their clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Hector R Perez, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, we have elected to not allow for data to be available to other researchers for secondary analyses.